CLINICAL TRIAL: NCT07010263
Title: A Multicenter, Randomized, Double-blind, Phase III Clinical Study of Comparing the Efficacy and Safety of AK112 (PD-1/VEGF Bispecific Antibody) Versus Placebo as Consolidation Treatment for Patients With Limited Stage Small-Cell Lung Cancer Who Have Not Progressed Following Concurrent Chemoradiation Therapy
Brief Title: A Study of AK112 as Consolidation Treatment for Patients With Limited Stage Small-cell Lung Cancer Who Have Not Progressed Following Concurrent Chemoradiation Therapy
Acronym: AK112-311
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK112-311
Record Dates: First submitted 2025-05-25; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Small Cell Lung Cancer
Keywords: AK112; Ivonescimab
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ak112 arm (Experimental): AK112 intravenous [IV]),every 3 weeks
  Interventions: Drug: AK112
- Placebo arm (Placebo Comparator): Placebo intravenous [IV]),every 3 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AK112 — AK112 20mg/kg, intravenous [IV]),Q3W
  Other Names: Ivonescimab
  Arms: Ak112 arm
Other: Placebo — Placebo, intravenous [IV]),Q3W
  Arms: Placebo arm

SUMMARY:
This is a randomized, double-blind, phase III clinical study to compare the efficacy and safety of AK112 to placebo as consolidation treatment for patients with limited stage small cell lung cancer who have not progressed following concurrent chemoradiation therapy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. The subjects voluntarily participated in the study with full informed consent and signed written informed consent form.
2. Aged ≥18 years on day fo signing the informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy ≥ 3 months
5. Histologically or cytologically confirmed small cell lung cancer.
6. Documented limited-stage SCLC (Stage I-III SCLC [T any, N any, M0] according to the American Joint Committee on Cancer Staging Manual [AJCC Cancer Staging Manual, 8th Edition] or the Veterans Administration Lung Study Group (VALG) stage.
7. Have Received concurrent chemoradiotherapy regimen as defined in protocol and have not progressed following concurrent chemoradiotherapy.
8. Adequate organ function.
9. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose and agree to take effective contraception measures during the study drug administration and within 120 days after the last dose.

Exclusion Criteria:

1. Histologically or cytological confirmed the presence of mixed small cell lung cancer or non-small cell lung cancer components.
2. Toxicities from previous anti-tumor treatments have not resolved to grade 0 or 1 based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0), or to the levels specified in inclusion/exclusion criteria, except for alopecia.
3. Symptoms or signs of primary disease deterioration that the investigator judges clinically unacceptable, such as cachexia.
4. Presence of pleural effusion, pericardial effusion, or ascites, which was clinically symptomatic or requiring frequent drainage.
5. History of active malignant tumors within the previous 5 years.
6. Received major surgery within 28 days prior to the first dose of study drug, or expected to undergo major surgery during the study period within 28 days after the first dose of study drug.
7. Uncontrolled comorbidities, including but not limited to decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis, and other related diseases..
8. Have serious neurological or mental illnesses, including dementia and epileptic seizures.
9. Pregnant or lactating women.
10. Have cardiovascular or cerebrovascular diseases or risk factors.
11. Prior treatments with systemic non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, etc.) within 2 weeks before the first administration of the study drugs. Prior treatment with Chinese herbal medicine or traditional Chinese patent medicines with anti-tumor indications within 1 weeks before the first administration of the study drugs.
12. Prior treatments targeting immune mechanisms, including, but not limited to, immune checkpoint inhibitors, immune checkpoint agonists, immune cell therapy.
13. Prior treatments with anti-angiogenic therapy.
14. Subjects requiring systemic treatment with corticosteroids (>10mg/day prednisone or equivalent dose) or other immunosuppressive drugs within 14 days prior to the first dose of study drug.
15. Known history of severe hypersensitivity reactions to other monoclonal antibodies or with a known history of allergy or hypersensitivity reactions to any of study drugs or their components.
16. Active autoimmune diseases that require systemic treatment within 2 years prior to the study, or autoimmune diseases that the investigator judges to be potentially recurrent or require planned treatment.
17. Known interstitial lung disease or non infectious pneumonia, which currently has symptoms or requires systemic corticosteroid treatment in the past,or investigator juges may affect the toxicity assessment or management related to the study treatment.
18. Known severe infection within 4 weeks prior to the first dose of study drug. Known active tuberculosis. Known active syphilis infection. Known history of immunodeficiency or positive HIV test results.
19. .Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
20. Active hepatitis B or active hepatitis C.
21. Received a live vaccine within 30 days prior to the first dose of study drug, or planning to receive a live vaccine during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-05-29 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival(PFS) assessed by Blinded independent center review(BIRC) | Approximately 6 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST v1.1

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 6 years
  OS is defined as the time from randomization or first dosing to death due to any cause.
PFS assessed by investigator per RECIST v1.1 | Approximately 6 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST v1.1
Objective Response Rate (ORR) assessed by BICR Per RECIST v1.1 | Approximately 6 years
ORR assessed by investigator Per RECIST v1.1 | Approximately 6 years
Disease control rate(DCR) assessed by BICR per RECIST v1.1 | Approximately 6 years
DCR assessed by investigator per RECIST v1.1 | Approximately 6 years
Duration of Response (DOR) assessed by BICR per RECIST v1.1 | Approximately 6 years
DOR assessed by investigator per RECIST v1.1 | Approximately 6 years
Number of participants with adverse event (AE) | Approximately 6 years
  The number of participants experiencing an AE and the severity of AEs will be assessed. AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Locations (40):
- China (40):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Longyan First Hospital, Longyan, Fujian
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Second Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jingzhou First People's Hospital, Jingzhou, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xuzhou Municipal Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Gannan Medical University, Gannan, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Ningxia Medical University General Hospital, Yinchuan, Ningxia
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Qingdao Central Hospital of Health and Rehabilitation Sciences University, Qingdao, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Sichuan People's Hospital, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Qujing First People's Hospital, Qujing, Yunnan
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang